CLINICAL TRIAL: NCT01138761
Title: Health Literacy for Children With Atopic Dermatitis and Their Caregivers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was significantly under target.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Gretchen K Carlisle, Research Scientist, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 1164097
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis
Keywords: pediatric atopic dermatitis; EASI; REALM-SF; nurse instruction; health literacy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Patient Education as Topic; Educational Status; Faculty, Nursing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physician/resident instruction (No Intervention): This arm is standard of care instruction given to parents/caregivers of children with atopic dermatitis by the dermatologist and/or dermatology resident during a patient visit.
- Nurse instruction (Active Comparator): Following the usual standard of care instruction by physician/resident (which both the treatment group and the non-treatment group will receive); the dermatology nurse will give enhanced instruction about skin care and medications to the caregivers/parents who were randomized to the treatment group.
  Interventions: Behavioral: Nurse instruction

INTERVENTIONS:
Behavioral: Nurse instruction — The dermatology nurse will give additional verbal and written instruction utilizing "teach-back" about skin care precautions and medication usage to the caregivers/parents in the "treatment" group.
  Other Names: patient education; caregiver instruction; teaching; medication compliance instruction; nurse teaching
  Arms: Nurse instruction

SUMMARY:
The purpose of this study is to determine the effectiveness of additional nursing instruction for the caregivers of newly diagnosed pediatric atopic dermatitis patients at the University of Missouri Dermatology clinic.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of additional nursing instruction for the caregivers of newly diagnosed pediatric atopic dermatitis patients at the University of Missouri Dermatology clinic. Caregivers of children with atopic dermatitis will be randomized to one of two instruction/education procedures. The goal is to determine if improved retention of information by caregivers/parents of children with atopic dermatitis is associated with better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New clinical diagnosis of pediatric atopic dermatitis, or existing atopic dermatitis but new patient to MU dermatology
* Age 7 or under

Exclusion Criteria:

* Age 8 or above

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Eczema Area and Severity Index (EASI) | EASI administered by blinded investigator at the initial visit, prior to teaching intervention; EASI again administered by same blinded investigator at visit 2 (at 4 weeks).
  The Eczema Area and Severity Index is used to document extent and severity of atopic dermatitis on child's skin at the beginning of the study and again at the follow-up visit. The purpose is to determine improvement or lack of improvement following teaching intervention by nurses in the dermatology clinic.

SECONDARY OUTCOMES:
Caregiver Questionnaire | Visit 2 (or Week 4 visit)
  A 27 item written questionnaire will be given to the parent/caregiver at visit 2. This questionnaire tests the retention of information given at visit 1 to subjects in both arms of the study (treatment and control group).

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Carlisle, MPH, Principal Investigator — University of Missouri, Columbia, MO; Jonathan A Dyer, MD, Principal Investigator — University of Missouri, Columbia, MO
Locations (1):
- University of Missouri Dermatology Clinic, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No